CLINICAL TRIAL: NCT07319949
Title: Evaluative Study on Predicting the Primary Site of Metastatic Tumors Using Transcriptomic Profiling for Tumor Tissue Origin Identification
Brief Title: Evaluating the Predictive Capability of Transcriptomic Profiling for Identifying the Primary Site of Metastatic Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of the Department of Breast Surgery, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: SRTCD-NO001
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Malignant Tumor With Metastasis; CUP
Keywords: Cancer of unknown primary; Specific RNA transcript; Tissue origin identification; Machine learning; Cancer diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be collected from patients who have been screened, enrolled, and have signed informed consent forms. Detectable sample types include fresh tissue samples, biopsy tissue samples, and formalin-fixed, paraffin-embedded (FFPE) tissue samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will enroll patients with metastatic malignancies. Tumor samples (fresh or formalin-fixed paraffin-embedded tissue specimens) will undergo RNA extraction and next-generation sequencing (RNA-seq). Once the raw data is obtained, the system will analyze the transcriptomic feature values (cancer-specific RNA transcripts and tissue-specific RNA transcripts) expressed in the tumor tissue samples to further predict tissue origin using a machine learning model. The output includes probabilities and confidence intervals for tissue origin.

DETAILED DESCRIPTION:
This is a non-interventional, observational study. Through a single-center, prospective clinical trial, the study aims to utilize the transcriptomic profiling for tumor tissue origin identification to predict the tissue origin of primary sites in metastatic tumors and evaluate the accuracy and specificity of this prediction solution.

Primary Endpoint:

The accuracy of the transcriptomic profiling for tumor tissue origin identification in predicting the primary site of metastatic tumors (expressed as overall accuracy with its 95% confidence interval).

Secondary Endpoints:

1. The specificity and sensitivity of the transcriptomic profiling for tumor tissue origin identification in predicting the primary site of metastatic tumors.
2. Exploratory analysis of characteristic molecular markers expressed in metastatic lesions from different primary sites.

ELIGIBILITY:
Inclusion Criteria

1. Clinically confirmed diagnosis of malignant tumor with metastasis;
2. Metastatic lesions confirmed as malignant by histopathology;
3. Sufficient surgical resection or biopsy specimens retained to meet the requirements for next-generation sequencing;
4. The participant (or their legal representative/guardian) has signed the informed consent form, confirming full understanding of the study's purpose and procedures, and voluntarily agrees to participate.

Exclusion Criteria:

1. The investigator deems the patient unable to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in Fudan University Shanghai Cancer Center, encompassing both outpatient and inpatient populations.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-10-13 (Estimated); Study Completion 2026-10-13 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the transcriptomic profiling for tumor tissue origin identification in predicting the primary site of metastatic tumors | through study completion, an average of 1 year
  Overall accuracy of the tumor tissue origin tracing transcriptome test for predicting the primary site of metastatic tumors (number of correct predictions/total evaluable cases); Specificity [true negatives/(true negatives + false positives)]; Sensitivity [true positives/(true positives + false negatives)].

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi Q, Li X, Liu Y, Chen Z, He X. FLIBase: a comprehensive repository of full-length isoforms across human cancers and tissues. Nucleic Acids Res. 2024 Jan 5;52(D1):D124-D133. doi: 10.1093/nar/gkad745. PMID 37697439
- [Background] Shi Q, Liu T, Hu W, Chen Z, He X, Li S. SRTdb: an omnibus for human tissue and cancer-specific RNA transcripts. Biomark Res. 2022 Apr 26;10(1):27. doi: 10.1186/s40364-022-00377-1. PMID 35473935
- [Background] Lee MS, Sanoff HK. Cancer of unknown primary. BMJ. 2020 Dec 7;371:m4050. doi: 10.1136/bmj.m4050. PMID 33288500